CLINICAL TRIAL: NCT00066430
Title: Infrared Coagulator For Treatment Of High Grade Squamous Intraepithelial Neoplasia (HSIL) in the Anal Canal In HIV Infected Individuals: A Pilot Study
Brief Title: Infrared Coagulation in Preventing Anal Cancer in Patients With HIV Who Have Anal Neoplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-032; CDR0000316109 (Other: NCI)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Anal Cancer; Precancerous Condition
Keywords: anal cancer; high-grade squamous intraepithelial lesion
MeSH Terms: conditions — Anus Neoplasms; Precancerous Conditions; Squamous Intraepithelial Lesions | interventions — Light Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infrared coagulator (Experimental)
  Interventions: Procedure: infrared photocoagulation therapy; Device: Infrared Coagulator

INTERVENTIONS:
Procedure: infrared photocoagulation therapy
Device: Infrared Coagulator — IRC treatment of up to 3 HGAIN lesions at baseline (study initiation). A second IRC treatment may be administered for recurrent lesions at the 3 month visit.
  Other Names: Redfield Infrared Coagulator (IRC) 2100

SUMMARY:
RATIONALE: Infrared coagulation may be effective in preventing the development of anal cancer in patients who have anal neoplasia.

PURPOSE: Pilot study to evaluate the effectiveness of infrared coagulation in preventing anal cancer in HIV-positive patients who have high-grade anal neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recurrence rate of high-grade squamous intraepithelial neoplasia in the anal canal of HIV-positive patients treated with infrared coagulation.
* Determine the time to recurrence and time to progression in patients treated with this procedure.
* Determine the toxicity of this procedure in these patients.
* Correlate CD4/CD8 count and HIV viral load with outcome in patients treated with this procedure.
* Correlate outcome with human papilloma virus subtype in patients treated with this procedure.

OUTLINE: This is an open-label, pilot, multicenter study.

Patients undergo treatment with an infrared coagulator in direct contact with the lesion for 1.5 seconds and necrotic tissue is then debrided. Treatment repeats to the level of the submucosal vessels under colposcopic guidance. A repeat biopsy is performed at 3 months to assess treatment success. Patients with incompletely treated lesions receive 1 more treatment. Up to 3 lesions are treated during each visit in the absence of disease progression or unacceptable toxicity.

Patients complete questionnaires regarding anal pain and discomfort at baseline, at 4 weeks, and at 3, 6, 9, and 12 months.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study within 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV positive
* Presence of internal anal lesions with histologically confirmed high-grade squamous intraepithelial neoplasia with at least 1 positive margin

  * No more than 3 lesions, each no more than 10 mm in diameter
* No evidence of microscopic invasion in any anal biopsy specimens
* No history of anal cancer

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Platelet count at least 50,000/mm^3
* CD4 count at least 50 cells/mm^3

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to lidocaine
* No anal insertions, including enemas or anal intercourse, for 24 hours before and at least 1 week after study treatment
* No prior severe photosensitivity reaction
* No active opportunistic infection
* No concurrent neoplasia requiring cytotoxic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Must be on stable regimen of highly active antiretroviral therapy (HAART) for at least 12 weeks prior to study entry unless CD4 count > 200/mm^3 AND no plans to initiate HAART within the next 3 months
* More than 14 days since prior acute treatment for an infection or other medical illness
* No prior infrared coagulation for anal dysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-09; Primary Completion 2004-09 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stier, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York